CLINICAL TRIAL: NCT02273414
Title: A Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Investigate the Safety, Tolerability, Biological Effects and Preliminary Pharmacokinetics of Increasing Repeated Oral Doses (9 Days Dosing) of BIIL 284 BS (Doses: 25 mg, 150 mg, 250 mg as WIF Tablets) in Healthy Male Volunteers
Brief Title: Study to Investigate the Safety, Tolerability, Biological Effects and Preliminary Pharmacokinetics of Increasing Doses of BIIL 284 BS in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 543.4
Record Dates: First submitted 2014-10-23; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (2):
- BIIL 284 BS - rising dose (Experimental)
  Interventions: Drug: BIIL 284 BS - rising dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIL 284 BS - rising dose
  Arms: BIIL 284 BS - rising dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of the present study is to obtain information about the safety and tolerability of BIIL 284 BS after repeated dosing, to find the pharmacologically active dose range by determination of the surrogate marker CD 11b (= Mac-1) and to obtain preliminary pharmacokinetic data concerning steady state and accumulation factor

ELIGIBILITY:
Inclusion Criteria:

* All participants are healthy males
* Age range from 21 to 50 years
* Broca-Index: within +- 20% of their normal weight
* In accordance with Good Clinical Practice (GCP) and local legislation each volunteer is supposed to give their written informed consent prior to admission to the study

Exclusion Criteria:

* Volunteers will be excluded from the study if the results of the medical examination or laboratory tests are judged by the clinical investigator to differ significantly from normal clinical values
* Volunteers with known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Volunteers with diseases of the central nervous system (such as epilepsy) or with psychiatric disorders
* Volunteers with history of orthostatic hypotension, fainting spells or blackouts
* Volunteers with chronic or relevant acute infections
* Volunteers with history of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Volunteers with eosinophilia > 7 %
* Volunteers who have taken a drug with a long half-life (>= 24 hours) within at least one month or less than ten half-lives of the respective drug before enrollment in the study
* Volunteers who received any drugs which might influence the results of the trial the week previous to the start of the study
* Volunteers who have participated in another study with an investigational drug within the last two months preceding this study
* Volunteers who smoke
* Volunteers who drink more than 60g of alcohol per day
* Volunteers who are dependent on drugs
* Volunteers who participated in excessive physical activities (e.g. competitive sports) within the last week before the study
* Volunteers who have donated blood within the last 4 weeks (>= 100 mL)

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 1999-07; Primary Completion 1999-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | up to 8 days after last drug administration
Number of subjects with abnormal changes in laboratory parameters | up to 8 days after last drug administration
Number of subjects with clinically significant changes in vital signs | up to 8 days after last drug administration
  Blood pressure, Pulse Rate, Respiratory Rate
Number of subjects with clinically significant changes in 12-lead electrocardiogram | up to 8 days after last drug administration

SECONDARY OUTCOMES:
AUC0-24h (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 24 hours) | up to 24 hours after drug administration
Cmax (Maximum measured concentration of the analyte in plasma) | up to 80 hours after drug administration
tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 80 hours after drug administration
t½ (Terminal half-life of the analyte in plasma) | up to 80 hours after drug administration
MRTtot (Total mean residence time) | up to 80 hours after drug administration
Vz/F (Apparent volume of distribution of the analyte during the terminal phase) | up to 80 hours after drug administration
CLtot/F (Total clearance after oral administration) | up to 80 hours after drug administration
Ae0-24h (Amount of analyte that is eliminated in urine from 0 to 24 hours) | up to 24 hours after drug administration
AUCss (Area under the plasma concentration-time curve at steady state) | up to 80 hours after drug administration
Cpre,ss (Predose concentration of the analyte in plasma at steady state) | up to 80 hours after drug administration
Changes in Leucotriene B4 (LTB4) induced Mac-1 expression | up to 24 hours after last treatment on day 9